CLINICAL TRIAL: NCT01489995
Title: A Randomized, Open-Label, 5-Period Crossover Study to Evaluate the Effect of Meal Type and Timing on the Pharmacokinetics of Migalastat Hydrochloride in Healthy Volunteers.
Brief Title: Migalastat Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116050
Record Dates: First submitted 2011-10-20; First posted 2011-12-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Fabry Disease
Keywords: Food effect; GR181413A; AT1001; migalastat hydrochloride; Lysosomal storage disorders; Pharmacokinetics
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases | interventions — migalastat; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Reference (Experimental): Fasted
  Interventions: Drug: A (migalastat)
- Glucose Drink (Experimental): Fed
  Interventions: Drug: B (migalastat)
- Before High Fat Meal (Experimental): Fed
  Interventions: Drug: C (migalastat)
- Before Light Meal (Experimental): Fed
  Interventions: Drug: D (migalastat)
- After Light Meal (Experimental): Fed
  Interventions: Drug: E (migalastat)

INTERVENTIONS:
Drug: A (migalastat) — 150 mg migalastat HCl in the fasting state (reference arm)
  Arms: Reference
Drug: B (migalastat) — 150 mg migalastat HCl with simultaneous consumption of a glucose drink
  Arms: Glucose Drink
Drug: C (migalastat) — 150 mg migalastat HCl 1 hour before consumption of a high fat meal
  Arms: Before High Fat Meal
Drug: D (migalastat) — 150 mg migalastat HCl 1 hour before consumption of a light meal
  Arms: Before Light Meal
Drug: E (migalastat) — 150 mg migalastat HCl 1 hour after consumption of a light meal
  Arms: After Light Meal

SUMMARY:
A 5-period crossover study to evaluate the effect of meal type and timing on migalastat HCl pharmacokinetics in healthy male and female subjects. Subjects will be randomly assigned to 1 of 5 treatment sequences and will receive each treatment over the course of 5 weekly periods.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, 5-period crossover study to evaluate the effect of meal type and timing on migalastat HCl pharmacokinetics in healthy male and female subjects between the ages of 18 and 65 years. A total of 20 subjects will be enrolled such that approximately 14 evaluable subjects complete dosing and critical assessments. Subjects will be randomly assigned to 1 of 5 treatment sequences and will receive each treatment over the course of 5 successive weekly periods including a single dose of migalastat HCl 150 mg in the fasting state as the reference treatment. There will be at least a 7-day washout period between each dose of migalastat HCl and a follow-up visit approximately 7 to 10 days after the last dose in Period 5.

All subjects will be screened within 28 days of admission to the clinical unit. In each period, subjects will check in to the clinical unit the day prior to drug administration and have relevant assessments to ensure continued eligibility for dose administration. On Day 1 of each period, subjects will receive a single dose of migalastat HCl within 1 of the following 5 treatment regimens as follows:

* 150 mg migalastat HCl in the fasting state (reference arm)
* 150 mg migalastat HCl with simultaneous consumption of a glucose drink
* 150 mg migalastat HCl 1 hour before consumption of a high fat meal
* 150 mg migalastat HCl 1 hour before consumption of a light meal
* 150 mg migalastat HCl 1 hour after consumption of a light meal

Subjects will be confined to the clinical unit for 24 hours after dosing with serial blood samples collected for PK analysis. Safety will be assessed throughout the study by monitoring clinical laboratory tests, ECGs, physical examinations, vital signs, and AEs.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 to 65 years inclusive
* Healthy, as determined by study physician
* Capable of giving informed consent

Exclusion Criteria:

* Positive for HIV or Hepatitis B and/or C viruses
* History of drug or alcohol abuse or addiction within 2 years
* Smoker or consumes tobacco products
* Participation in a clinical trial within 30 days of scheduled first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of migalastat HCl after a single dose | 5 weeks (60 PK timepoints)
  Cmax
Time of occurence of maximum observed plasma concentration of migalastat HCl after a single dose | 5 weeks (60 PK timepoints)
  tmax
Area under the plasma concentration-time curve of migalastat HCl after a single dose from time 0 (before dosing) to infinity | 5 weeks (60 PK timepoints)
  AUC (0 to infinity)
Terminal phase half life of migalastat HCl after a single dose | 5 weeks (60 PK timepoints)
  t1/2
Apparent clearance following oral dosing of migalastat HCl after a single dose | 5 weeks (60 PK timepoints)
  CL/F
Area under the plasma concentration-time curve of migalastat HCl after a single dose from time 0 (before dosing) to the time of the last quantifiable concentration | 5 weeks (60 PK timepoints)
  AUC (0 to t)

SECONDARY OUTCOMES:
Adverse Events | 5 weeks
Clinical Laboratory Tests | 5 weeks
Vital Signs | 5 weeks
ECGs | 5 weeks
Physical Examination | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — AmicusTherapeutics
Locations (1):
- GSK Investigational Site, Austin, Texas, United States